CLINICAL TRIAL: NCT02910557
Title: A Postmarketing Prospective Cohort Study of Melanoma Patients Treated With IMLYGIC® in Clinical Practice to Characterize Risk of Herpetic Infection Among Patients, Close Contacts, Health Care Providers & Long-term Safety in Treated Patients
Brief Title: Postmarketing Prospective Study of Melanoma Patients Treated With IMLYGIC® to Characterize Risk of Herpetic Infection
Status: Completed | Type: Observational
Sponsor: Amgen (Industry)
Responsible Party: Sponsor
Other Study IDs: 20130193
Record Dates: First submitted 2016-09-07; First posted 2016-09-22 (Estimated); Last update posted 2026-02-05 (Actual); Status verified 2026-02

CONDITIONS: Melanoma; Herpetic Infection
Keywords: IMLYGIC; Talimogene Laherparepvec; Herpetic; Infection Melanoma
MeSH Terms: conditions — Melanoma

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
A postmarketing Cohort study of Melanoma patients treated with IMLYGIC (Talimogene Laherparepvec) in clinical Practice to Characterize the risk of herpetic infection with detection of Talimogene Laherparepvec DNA among patients, close contacts, and health care providers; and long term safety in treated patients for up to 5 years after the first IMLYGIC dose.

ELIGIBILITY:
Inclusion Criteria:

* Patient has provided written informed consent
* Patient is an adult (≥ 18 years of age at the time of informed consent) with a diagnosis of melanoma
* Patient enrolled within 1 month of receiving the first dose of IMLYGIC for the treatment of melanoma

Exclusion Criteria:

- Patient has a prior history of being a subject in an interventional clinical trial for IMLYGIC

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: This postmarketing prospective cohort study will follow melanoma patients for up to 5 years after the first IMLYGIC dose in clinical practice. There is no experimental intervention, and the study population will receive standard-of-care treatment as determined by their treating physician.
Sampling Method: Non-Probability Sample
Enrollment: 187 (Actual)
Dates: Start 2017-08-10 (Actual); Primary Completion 2026-01-30 (Actual); Study Completion 2026-01-30 (Actual)

PRIMARY OUTCOMES:
Incidence Rate | Up to 5 years
  Estimate the incidence rate of herpetic infection with detection of talimogene laherparepvec (T-VEC) DNA among patients for up to 5 years after the first IMLYGIC dose.

SECONDARY OUTCOMES:
Herpectic Infection with T-VEC DNA for Close Contacts and Healthcare Providers (HCPs) | Through study completion, average of 5 years
  Count the number of herpetic infections with detection of T-VEC DNA among close contacts and HCPs.
Incidence of Herpetic Infection with T-VEC in Patients During Treatment | Through treatment period, up to 1 year
  Estimate the incidence rate of herpetic infection with detection of T-VEC DNA among patients during treatment with IMLYGIC.
Incidence of Herpetic Infection with T-VEC in Patients After Treatment | Through study completion, average of 5 years
  Estimate the incidence rate of herpetic infection with detection of T-VEC DNA among patients after discontinuation of IMLYGIC.
Incidence of Herpes Simplex Virus 1 (HSV-1) DNA in Patients During Treatment | Through treatment period, up to 1 year
  Estimate the incidence rate of herpetic infection with detection of wild-type HSV-1 DNA among patients during treatment with IMLYGIC.
Incidence of HSV-1 DNA in Patients After Treatment | Through study completion, average of 5 years
  Estimate the incidence rate of herpetic infection with detection of wild-type HSV-1 DNA among patients after discontinuation of IMLYGIC.
Patient Demographics | Through study completion, average of 5 years
  The following baseline variables will be recorded: sex, age, Eastern Cooperative Oncology Group (ECOG) performance status.
Use of Drug Therapies | Through study completion, average of 5 years
  Describe the use of IMLYGIC, other anti-cancer therapy, anti-herpetic therapy.
Incidence of Adverse Events and Serious Adverse Events in Patients | Through study completion, average of 5 years
  Incidence of adverse events and serious adverse events during and after treatment with IMLYGIC
Overall Survival | Through study completion, average of 5 years
  Survival is defined by the time to death from the date of the first use of IMLYGIC.

CONTACTS AND LOCATIONS:
Overall Officials: MD, Study Director — Amgen
Locations (23):
- United States (9):
  - Corazon United States of America, LLC doing business as Life Clinical Trials, Coral Springs, Florida
  - Mercy Medical Center, Baltimore, Maryland
  - Jefferson City Medical Group PC, Jefferson City, Missouri
  - TriHealth Cancer Institute - Kenwood, Cincinnati, Ohio
  - University of Pittsburgh Medical Center, Pittsburgh, Pennsylvania
  - Allegheny Health Network, Pittsburgh, Pennsylvania
  - University of Tennessee Medical Center, Knoxville, Tennessee
  - Intermountain Medical Center, Murray, Utah
  - University of Wisconsin Hospital and Clinics, Madison, Wisconsin
- Austria (4):
  - Medizinische Universitaet Graz, Graz
  - Ordensklinikum Linz Elisabethinen, Linz
  - Landeskrankenhaus Salzburg, Salzburg
  - Universitaetsklinikum Sankt Poelten, Sankt Pölten
- Israel (2):
  - Rambam Medical Center, Haifa
  - Sheba Medical Center, Ramat Gan
- Switzerland (3):
  - Universitaetsspital Basel, Basel
  - Kantonsspital Graubuenden, Chur
  - Universitaetsspital Zuerich, Zuerich Flughafen
- United Kingdom (5):
  - Cheltenham General Hospital, Cheltenham
  - Guys Hospital, London
  - Royal Marsden Hospital, London
  - Churchill Hospital, Oxford
  - Musgrove Park Hospital, Taunton

IPD SHARING:
Plan to Share IPD: Yes
De-identified individual patient data for variables necessary to address the specific research question in an approved data sharing request
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: Data sharing requests relating to this study will be considered beginning 18 months after the study has ended and either 1) the product and indication (or other new use) have been granted marketing authorization in both the US and Europe or 2) clinical development for the product and/or indication discontinues and the data will not be submitted to regulatory authorities. There is no end date for eligibility to submit a data sharing request for this study.
Access Criteria: Qualified researchers may submit a request containing the research objectives, the Amgen product(s) and Amgen study/studies in scope, endpoints/outcomes of interest, statistical analysis plan, data requirements, publication plan, and qualifications of the researcher(s). In general, Amgen does not grant external requests for individual patient data for the purpose of re-evaluating safety and efficacy issues already addressed in the product labelling. Requests are reviewed by a committee of internal advisors, and if not approved, may be further arbitrated by a Data Sharing Independent Review Panel. Upon approval, information necessary to address the research question will be provided under the terms of a data sharing agreement. This may include anonymized individual patient data and/or available supporting documents, containing fragments of analysis code where provided in analysis specifications. Further details are available at the link below.
URL: https://www.amgen.com/datasharing

REFERENCES:
- See also: AmgenTrials clinical trials website — http://www.amgentrials.com